CLINICAL TRIAL: NCT00208325
Title: Clinical Evaluation of the P.F.C. Sigma (Fixed Bearing) and P.F.C. Sigma RP (Mobile Bearing) Total Knee Systems
Brief Title: PFC Sigma Fixed and Mobile Knee Study
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: The study was terminated at the point the primary endpoint and early milestones were reached and because long term outcomes were available from other sources
Sponsor: DePuy International (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: CT 9923
Record Dates: First submitted 2005-09-13; First posted 2005-09-21 (Estimated); Results first posted 2016-07-20 (Estimated); Last update posted 2016-09-13 (Estimated); Status verified 2016-08

CONDITIONS: Osteoarthritis, Knee
MeSH Terms: conditions — Osteoarthritis, Knee

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (4):
- PFC Sigma Fixed Bearing PCL Sacrificed (Other): PFC Sigma Fixed Bearing Total Knee System with PCL Sacrificed
  Interventions: Device: P.F.C Sigma Fixed Bearing total knee system
- PFC Sigma RP PCL Sacrificed (Active Comparator): PFC Sigma Rotating Platform Total Knee System with PCL Sacrificed
  Interventions: Device: P.F.C Sigma RP Mobile Bearing knee system
- PFC Sigma Fixed Bearing PCL Retained (Other): PFC Sigma Fixed Bearing Total Knee System with PCL Retained
  Interventions: Device: P.F.C Sigma Fixed Bearing total knee system
- PFC Sigma RP PCL Retained (Active Comparator): PFC Sigma Rotating Platform Total Knee System with PCL Retained
  Interventions: Device: P.F.C Sigma RP Mobile Bearing knee system

INTERVENTIONS:
Device: P.F.C Sigma Fixed Bearing total knee system — Orthopaedic implant for total knee replacement
  Arms: PFC Sigma Fixed Bearing PCL Retained; PFC Sigma Fixed Bearing PCL Sacrificed
Device: P.F.C Sigma RP Mobile Bearing knee system — Orthopaedic implant for total knee replacement
  Arms: PFC Sigma RP PCL Retained; PFC Sigma RP PCL Sacrificed

SUMMARY:
The primary objective of this investigation is to evaluate the performance (in terms of post-operative active range of motion at one year) of the P.F.C. Sigma and P.F.C. Sigma Rotating Platform total knee systems in clinical practice.

DETAILED DESCRIPTION:
The secondary objectives of this investigation are:To evaluate the performance of the P.F.C. Sigma and P.F.C. Sigma Rotating Platform total knee systems in clinical practice. To evaluate the impact of patellar resurfacing on the performance of the P.F.C. Sigma and the P.F.C. Sigma Rotating Platform total knee systems. To evaluate the impact of Posterior Cruciate Ligament (PCL) sacrifice or retention on the performance of the P.F.C. Sigma and the P.F.C. Sigma Rotating Platform total knee systems.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female subjects may be recruited to the evaluation.
2. Age - there are no restrictions relating to age of the patient. The patient's age must be considered suitable by the clinical investigator for a bi-compartmental or tri-compartmental knee arthroplasty using either of the two systems available in the evaluation.
3. Subjects who are able to give voluntary, written informed consent to participate in this investigation and from whom consent has been obtained.
4. Subjects who, in the opinion of the Investigator, are able to understand this investigation, co-operate with the investigational procedures and are willing to return to the hospital for all the required post-operative follow-ups.
5. Subjects who require a bi-compartmental or tri-compartmental knee arthroplasty for primary surgical management of idiopathic osteoarthritis.
6. Patients who in the opinion of the Clinical Investigator are considered to be suitable for treatment with a fixed or mobile bearing knee system and who are suitable for patella resurfacing.

Exclusion Criteria:

1. Patients who, in the opinion of the Investigator, have an existing condition that would compromise their participation and follow-up in this study.
2. Patients who require revision total knee arthroplasty surgery.
3. Patients with any tibial deformity requiring tibial component augmentation.
4. Patients whom, in the opinion of the Clinical Investigator, require a constrained prosthesis.
5. Patients with Rheumatoid Arthritis.
6. Patients with a pathology which, in the opinion of the Clinical Investigator, will adversely affect healing.
7. Patients with other disorders which, in the opinion of the Clinical Investigator, will / could impair rehabilitation.
8. Contra-indications for use of the device, as detailed in the package insert.
9. Women who are pregnant.
10. Subjects who are known drug or alcohol abusers or with psychological disorders that could effect follow-up care or treatment outcomes.
11. Subjects who are currently involved in another clinical study with an investigational product.
12. Subjects who are currently involved in any injury litigation claims.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 754 (Actual)
Dates: Start 2000-05; Primary Completion 2009-01 (Actual); Study Completion 2010-09 (Actual)

CONTACTS AND LOCATIONS:
Locations (4):
- United Kingdom (4):
  - Glasgow Royal Infirmary, Glasgow
  - Glasgow Western Infirmary, Glasgow
  - Northampton General Hospital, Northampton
  - Nottingham City Hospital, Nottingham

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 754 subjects were consented into the study, however only 720 received study treatment.
Groups:
- PFC Fixed Bearing PCL Sacrificed; PFC Fixed Bearing PCL Retained: Fixed bearing
  P.F.C Sigma Fixed Bearing Total knee system: Orthopaedic implant for total knee replacement
- PFC Mobile Bearing PCL Sacrificed: Mobile bearing
  P.F.C Sigma RP Mobile Bearing knee system: Orthopaedic implant for total knee replacement
- PFC Mobile Bearing PCL Retained: Mobile bearing
  P.F.C Sigma Mobile Bearing Total knee system: Orthopaedic implant for total knee replacement
Period: Overall Study
Arm/Group | PFC Fixed Bearing PCL Sacrificed | PFC Mobile Bearing PCL Sacrificed | PFC Fixed Bearing PCL Retained | PFC Mobile Bearing PCL Retained
Started | 193 | 196 | 170 | 161
Completed | 142 | 142 | 156 | 147
Not Completed | 51 | 54 | 14 | 14
Not completed — Death | 18 | 19 | 7 | 5
Not completed — Withdrawal by Subject | 0 | 1 | 0 | 0
Not completed — Revision | 4 | 1 | 0 | 4
Not completed — Lost to Follow-up | 1 | 0 | 2 | 0
Not completed — Unsurfaced to Resurfaced Patella | 4 | 4 | 1 | 3
Not completed — Does not wish to Continue in Study | 5 | 8 | 3 | 2
Not completed — Other | 2 | 1 | 1 | 0
Not completed — Mis-Randomized | 17 | 20 | 0 | 0

BASELINE CHARACTERISTICS:
Population: All participants who received treatment and were not mis-randomized.
Groups:
- PFC Fixed Bearing PCL Sacrificed: PFC Sigma Fixed Bearing Total Knee System with PCL Sacrificed
  P.F.C Sigma Fixed Bearing total knee system: Orthopaedic implant for total knee replacement
- Total: Total of all reporting groups
Arm/Group | PFC Fixed Bearing PCL Sacrificed | PFC Sigma RP PCL Sacrificed | PFC Sigma Fixed Bearing PCL Retained | PFC Sigma RP PCL Retained | Total
Number analyzed (Participants) | 176 | 176 | 170 | 161 | 683
Age, Continuous [Mean (Standard Deviation); unit: years] | 69.8 (8.16) | 70.2 (7.60) | 70.1 (7.88) | 69.2 (8.59) | 69.8 (8.06)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 94 | 96 | 102 | 87 | 379
  Male | 82 | 80 | 68 | 74 | 304
Region of Enrollment [Number; unit: participants]
  United Kingdom | 176 | 176 | 170 | 161 | 683

OUTCOME MEASURES:

1. Primary Outcome: To Compare Range of Motion Between Sigma RP and Sigma Fixed Treatment Groups in PCL Sacrificing Arm
Description: Range of motion is knee flexion (how far the patient can bend their knee) minus knee extension (how far the patient can straighten their knee). The result of this subtraction is the range of motion (bending and straightening) for that knee.
Time Frame: 1 year
Population: Due to consent withdrawals, deaths, lost to follow up, revisions, subjects whose patella were resurfaced, mis-randomized, those who did not wish to continue in the study, and incomplete or unavailable assessments, 168 subjects in the PFC Sigma Fixed Bearing and 167 subjects in the PFC Sigma RP Treatment Groups were available for this outcome.
Measure: Mean (Standard Deviation); unit: degrees
Arm/Group | PFC Fixed Bearing PCL Sacrificed | PFC Sigma RP PCL Sacrificed
Number analyzed (Participants) | 168 | 167
degrees | 108.8 (13.41) | 108.4 (12.54)

2. Primary Outcome: To Compare Range of Motion Between Sigma RP and Sigma Fixed Treatment Groups in PCL Retaining Arm
Description: as for outcome 1
Time Frame: 1 year
Population: Due to consent withdrawals, deaths, lost to follow up, revisions, subjects whose patella were resurfaced, mis-randomized, those who did not wish to continue in the study, and incomplete or unavailable assessments, 158 subjects in the PFC Sigma Fixed Bearing and 155 subjects in the PFC Sigma RP Treatment Groups were available for this outcome.
Measure: Mean (Standard Deviation); unit: degrees
Arm/Group | PFC Sigma Fixed Bearing PCL Retained | PFC Sigma RP PCL Retained
Number analyzed (Participants) | 158 | 155
degrees | 100.6 (12.94) | 101.6 (12.24)

3. Primary Outcome: To Compare the Change in Range of Motion From Pre-op to 1 Year Between Sigma RP and Sigma Fixed Treatment Groups in PCL Sacrificing Arm
Description: as for outcome 1
Time Frame: Change from pre-op to 1 year
Population: Due to consent withdrawals, deaths, lost to follow up, revisions, subjects whose patella were resurfaced, mis-randomized, those who did not wish to continue in the study, and incomplete or unavailable assessments, 164 subjects in the PFC Sigma Fixed Bearing and 164 subjects in the PFC Sigma RP Treatment Groups were available for this outcome.
Measure: Mean (Standard Deviation); unit: degrees
Arm/Group | PFC Fixed Bearing PCL Sacrificed | PFC Sigma RP PCL Sacrificed
Number analyzed (Participants) | 164 | 164
degrees | 13.4 (17.17) | 12.3 (18.70)

4. Primary Outcome: To Compare the Change in Range of Motion From Pre-op to 1 Year Between Sigma RP and Sigma Fixed Treatment Groups in PCL Retaining Arm
Description: as for outcome 1
Time Frame: Change from pre-op to 1 year
Population: Due to consent withdrawals, deaths, lost to follow up, revisions, subjects whose patella were resurfaced, mis-randomized, those who did not wish to continue in the study, and incomplete or unavailable assessments, 158 subjects in the PFC Sigma Fixed Bearing and 153 subjects in the PFC Sigma RP Treatment Groups were available for this outcome.
Measure: Mean (Standard Deviation); unit: degrees
Arm/Group | PFC Sigma Fixed Bearing PCL Retained | PFC Sigma RP PCL Retained
Number analyzed (Participants) | 158 | 153
degrees | 5.8 (15.83) | 8.1 (15.74)

5. Secondary Outcome: To Compare the Change in Range of Motion From Pre-op to 2 Years Between Sigma RP and Sigma Fixed Treatment Groups in PCL Sacrificing Arm
Description: as for outcome 1
Time Frame: Change from pre-op to 2 years
Population: Due to consent withdrawals, deaths, lost to follow up, revisions, subjects whose patella were resurfaced, mis-randomized, those who did not wish to continue in the study, and incomplete or unavailable assessments, 156 subjects in the PFC Sigma Fixed Bearing and 148 subjects in the PFC Sigma RP Treatment Groups were available for this outcome.
Measure: Mean (Standard Deviation); unit: degrees
Arm/Group | PFC Fixed Bearing PCL Sacrificed | PFC Sigma RP PCL Sacrificed
Number analyzed (Participants) | 156 | 148
degrees | 13.9 (15.81) | 12.0 (17.99)

6. Secondary Outcome: To Compare the Change in Range of Motion From Pre-op to 2 Years Between Sigma RP and Sigma Fixed Treatment Groups in PCL Retaining Arm
Description: as for outcome 1
Time Frame: Change from pre-op to 2 years
Population: Due to consent withdrawals, deaths, lost to follow up, revisions, subjects whose patella were resurfaced, mis-randomized, those who did not wish to continue in the study, and incomplete or unavailable assessments, 170 subjects in the PFC Sigma Fixed Bearing and 161 subjects in the PFC Sigma RP Treatment Groups were available for this outcome.
Measure: Mean (Standard Deviation); unit: degrees
Arm/Group | PFC Sigma Fixed Bearing PCL Retained | PFC Sigma RP PCL Retained
Number analyzed (Participants) | 170 | 161
degrees | 8.7 (14.74) | 10.2 (15.72)

7. Secondary Outcome: To Compare the Change in Range of Motion From Pre-op to 5 Years Between Sigma RP and Sigma Fixed Treatment Groups in PCL Sacrificing Arm
Description: as for outcome 1
Time Frame: Change from pre-op to 5 years
Population: Due to consent withdrawals, deaths, lost to follow up, revisions, subjects whose patella were resurfaced, mis-randomized, those who did not wish to continue in the study, and incomplete or unavailable assessments, 123 subjects in the PFC Sigma Fixed Bearing and 124 subjects in the PFC Sigma RP Treatment Groups were available for this outcome.
Measure: Mean (Standard Deviation); unit: degrees
Arm/Group | PFC Fixed Bearing PCL Sacrificed | PFC Sigma RP PCL Sacrificed
Number analyzed (Participants) | 123 | 124
degrees | 15.2 (15.46) | 14.5 (18.77)

8. Secondary Outcome: To Compare the Change in Oxford Knee Score From Pre-op to 2 Years Between Sigma RP and Sigma Fixed Treatment Groups in PCL Retaining Arm
Description: The Oxford Knee Score (OKS) is a 12 to 60 point patient reported outcome (PRO) score (where 12 indicates the best outcome) that evaluates the affected knee. The total score is composed of Pain and Function.
Time Frame: Change from pre-op to 2 years
Population: Due to consent withdrawals, deaths, lost to follow up, revisions, subjects whose patella were resurfaced, mis-randomized, those who did not wish to continue in the study, and incomplete or unavailable assessments, 145 subjects in the PFC Sigma Fixed Bearing and 138 subjects in the PFC Sigma RP Treatment Groups were available for this outcome.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | PFC Sigma Fixed Bearing PCL Retained | PFC Sigma RP PCL Retained
Number analyzed (Participants) | 145 | 138
units on a scale | -19.1 (8.35) | -17.6 (9.92)

9. Secondary Outcome: To Compare the Change in Oxford Knee Score From Pre-op to 2 Years Between Sigma RP and Sigma Fixed Treatment Groups in PCL Sacrificing Arm
Description: as for outcome 8
Time Frame: Change from pre-op to 2 years
Population: Due to consent withdrawals, deaths, lost to follow up, revisions, subjects whose patella were resurfaced, mis-randomized, those who did not wish to continue in the study, and incomplete or unavailable assessments, 134 subjects in the PFC Sigma Fixed Bearing and 118 subjects in the PFC Sigma RP Treatment Groups were available for this outcome.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | PFC Fixed Bearing PCL Sacrificed | PFC Sigma RP PCL Sacrificed
Number analyzed (Participants) | 134 | 118
units on a scale | -18.8 (9.93) | -18.1 (8.90)

10. Secondary Outcome: To Compare the Change in Oxford Knee Score From Pre-op to 5 Years Between Sigma RP and Sigma Fixed Treatment Groups in PCL Sacrificing Arm
Description: as for outcome 8
Time Frame: Change from pre-op to 5 years
Population: Due to consent withdrawals, deaths, lost to follow up, revisions, subjects whose patella were resurfaced, mis-randomized, those who did not wish to continue in the study, and incomplete or unavailable assessments, 114 subjects in the PFC Sigma Fixed Bearing and 111 subjects in the PFC Sigma RP Treatment Groups were available for this outcome.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | PFC Fixed Bearing PCL Sacrificed | PFC Sigma RP PCL Sacrificed
Number analyzed (Participants) | 114 | 111
units on a scale | -20.4 (10.33) | -19.9 (8.95)

11. Secondary Outcome: To Compare the Change in American Knee Society Knee Score From Pre-op to 2 Years Between Sigma RP and Sigma Fixed Treatment Groups in PCL Sacrificing Arm
Description: American Knee Society (AKS) knee score is a 0-100 point score (where 100 indicates excellent knee condition) that evaluates the affected knee. The knee score is composed of Pain, Range of Motion, and Stability.
Time Frame: Change from pre-op to 2 years
Population: Due to consent withdrawals, deaths, lost to follow up, revisions, subjects whose patella were resurfaced, mis-randomized, those who did not wish to continue in the study, and incomplete or unavailable assessments, 154 subjects in the PFC Sigma Fixed Bearing and 143 subjects in the PFC Sigma RP Treatment Groups were available for this outcome.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | PFC Fixed Bearing PCL Sacrificed | PFC Sigma RP PCL Sacrificed
Number analyzed (Participants) | 154 | 143
units on a scale | 57.2 (18.66) | 56.8 (18.09)

12. Secondary Outcome: To Compare the Change in American Knee Society Knee Score From Pre-op to 2 Years Between Sigma RP and Sigma Fixed Treatment Groups in PCL Retaining Arm
Description: as for outcome 11
Time Frame: Change from pre-op to 2 years
Population: Due to consent withdrawals, deaths, lost to follow up, revisions, subjects whose patella were resurfaced, mis-randomized, those who did not wish to continue in the study, and incomplete or unavailable assessments, 152 subjects in the PFC Sigma Fixed Bearing and 143 subjects in the PFC Sigma RP Treatment Groups were available for this outcome.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | PFC Sigma Fixed Bearing PCL Retained | PFC Sigma RP PCL Retained
Number analyzed (Participants) | 152 | 143
units on a scale | 50.7 (21.02) | 49.5 (24.67)

13. Secondary Outcome: To Compare the Change in American Knee Society Knee Score From Pre-op to 5 Years Between Sigma RP and Sigma Fixed Treatment Groups in PCL Sacrificing Arm
Description: as for outcome 11
Time Frame: Change from pre-op to 5 years
Population: Due to consent withdrawals, deaths, lost to follow up, revisions, subjects whose patella were resurfaced, mis-randomized, those who did not wish to continue in the study, and incomplete or unavailable assessments, 122 subjects in the PFC Sigma Fixed Bearing and 120 subjects in the PFC Sigma RP Treatment Groups were available for this outcome.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | PFC Fixed Bearing PCL Sacrificed | PFC Sigma RP PCL Sacrificed
Number analyzed (Participants) | 122 | 120
units on a scale | 57.9 (19.42) | 55.6 (20.36)

14. Secondary Outcome: To Compare the Change in American Knee Society Function Score From Pre-op to 2 Years Between Sigma RP and Sigma Fixed Treatment Groups in PCL Sacrificing Arm
Description: American Knee Society (AKS) function score is a 0-100 point score (where 100 indicates excellent knee function) that evaluates the affected knee. The function score is composed of walking and stair climbing ability.
Time Frame: Change from pre-op to 2 years
Population: Due to consent withdrawals, deaths, lost to follow up, revisions, subjects whose patella were resurfaced, mis-randomized, those who did not wish to continue in the study, and incomplete or unavailable assessments, 155 subjects in the PFC Sigma Fixed Bearing and 144 subjects in the PFC Sigma RP Treatment Groups were available for this outcome.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | PFC Fixed Bearing PCL Sacrificed | PFC Sigma RP PCL Sacrificed
Number analyzed (Participants) | 155 | 144
units on a scale | 23.8 (22.18) | 26.1 (21.47)

15. Secondary Outcome: To Compare the Change in American Knee Society Function Score From Pre-op to 2 Years Between Sigma RP and Sigma Fixed Treatment Groups in PCL Retaining Arm
Description: as for outcome 14
Time Frame: Change from pre-op to 2 years
Population: Due to consent withdrawals, deaths, lost to follow up, revisions, subjects whose patella were resurfaced, mis-randomized, those who did not wish to continue in the study, and incomplete or unavailable assessments, 154 subjects in the PFC Sigma Fixed Bearing and 146 subjects in the PFC Sigma RP Treatment Groups were available for this outcome.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | PFC Sigma Fixed Bearing PCL Retained | PFC Sigma RP PCL Retained
Number analyzed (Participants) | 154 | 146
units on a scale | 25.0 (22.51) | 23.6 (19.62)

16. Secondary Outcome: To Compare the Change in American Knee Society Function Score From Pre-op to 5 Years Between Sigma RP and Sigma Fixed Treatment Groups in PCL Sacrificing Arm
Description: as for outcome 14
Time Frame: Change from pre-op to 5 years
Population: Due to consent withdrawals, deaths, lost to follow up, revisions, subjects whose patella were resurfaced, mis-randomized, those who did not wish to continue in the study, and incomplete or unavailable assessments, 124 subjects in the PFC Sigma Fixed Bearing and 125 subjects in the PFC Sigma RP Treatment Groups were available for this outcome.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | PFC Fixed Bearing PCL Sacrificed | PFC Sigma RP PCL Sacrificed
Number analyzed (Participants) | 124 | 125
units on a scale | 20.3 (24.54) | 20.5 (22.06)

17. Secondary Outcome: To Compare the Percentage of Subjects With No Anterior Knee Pain Between Sigma RP and Sigma Fixed Treatment Groups in PCL Sacrificing Arm
Description: Anterior Knee Pain is assessed by the patient into 1 of 4 categories: None, Mild, Moderate, or Severe. The percentage of participants with no anterior knee pain is reported in the data table.
Time Frame: 2 years
Population: Due to consent withdrawals, deaths, lost to follow up, revisions, subjects whose patella were resurfaced, mis-randomized, those who did not wish to continue in the study, and incomplete or unavailable assessments, 176 subjects in the PFC Sigma Fixed Bearing and 176 subjects in the PFC Sigma RP Treatment Groups were available for this outcome.
Measure: Number; unit: percentage of participants
Arm/Group | PFC Fixed Bearing PCL Sacrificed | PFC Sigma RP PCL Sacrificed
Number analyzed (Participants) | 176 | 176
percentage of participants | 73 | 67

18. Secondary Outcome: To Compare the Percentage of Subjects With No Anterior Knee Pain Between Sigma RP and Sigma Fixed Treatment Groups in PCL Retaining Arm
Description: as for outcome 17
Time Frame: 2 years
Population: as for outcome 6
Measure: Number; unit: percentage of participants
Arm/Group | PFC Sigma Fixed Bearing PCL Retained | PFC Sigma RP PCL Retained
Number analyzed (Participants) | 170 | 161
percentage of participants | 76 | 76

19. Secondary Outcome: To Compare the Percentage of Subjects With No Anterior Knee Pain Between Sigma RP and Sigma Fixed Treatment Groups in PCL Sacrificing Arm
Description: as for outcome 17
Time Frame: 5 Years
Population: as for outcome 17
Measure: Number; unit: percentage of participants
Arm/Group | PFC Fixed Bearing PCL Sacrificed | PFC Sigma RP PCL Sacrificed
Number analyzed (Participants) | 176 | 176
percentage of participants | 61 | 53

20. Secondary Outcome: To Compare the Percentage of Subjects With Good Quadriceps Strength Between Sigma RP and Sigma Fixed Treatment Groups in PCL Sacrificing Arm
Description: Quadriceps Strength is assessed by the patient into 1 of 3 categories: Good, Fair, or Poor. The percentage of participants with good quadriceps strength is reported in the data table.
Time Frame: 2 years
Population: as for outcome 17
Measure: Number; unit: percentage of participants
Arm/Group | PFC Fixed Bearing PCL Sacrificed | PFC Sigma RP PCL Sacrificed
Number analyzed (Participants) | 176 | 176
percentage of participants | 88 | 85

21. Secondary Outcome: To Compare the Percentage of Subjects With Good Quadriceps Strength Between Sigma RP and Sigma Fixed Treatment Groups in PCL Retaining Arm
Description: as for outcome 20
Time Frame: 2 years
Population: as for outcome 6
Measure: Number; unit: percentage of participants
Arm/Group | PFC Sigma Fixed Bearing PCL Retained | PFC Sigma RP PCL Retained
Number analyzed (Participants) | 170 | 161
percentage of participants | 81 | 82

22. Secondary Outcome: To Compare the Percentage of Subjects With Good Quadriceps Strength Between Sigma RP and Sigma Fixed Treatment Groups in PCL Sacrificing Arm
Description: as for outcome 20
Time Frame: 5 Years
Population: as for outcome 17
Measure: Number; unit: percentage of participants
Arm/Group | PFC Fixed Bearing PCL Sacrificed | PFC Sigma RP PCL Sacrificed
Number analyzed (Participants) | 176 | 176
percentage of participants | 65 | 68

23. Secondary Outcome: To Compare the Change in SF-12 Physical Health Score From Pre-op to 2 Years Between Sigma RP and Sigma Fixed Treatment Groups in PCL Sacrificing Arm
Description: The 12-Item Short Form Health Survey (SF-12) is a patient reported outcome survey that represents overall subjective health status by measuring eight health-related parameters (each scored from 0 [poor health] to 100 [better health]): body pain, general mental health, perception of general health, physical functioning, role limitations caused by mental condition, role limitations caused by a physical condition, social functioning, and vitality. The survey is converted into 2 summary measures that are scored from 0 to 100 (where 100 indicates the highest level of health) - the Physical Component Score (PCS-12) and Mental Component Score (MCS-12).
Time Frame: Change from pre-op to 2 years
Population: Due to consent withdrawals, deaths, lost to follow up, revisions, subjects whose patella were resurfaced, mis-randomized, those who did not wish to continue in the study, and incomplete or unavailable assessments, 130 subjects in the PFC Sigma Fixed Bearing and 118 subjects in the PFC Sigma RP Treatment Groups were available for this outcome.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | PFC Fixed Bearing PCL Sacrificed | PFC Sigma RP PCL Sacrificed
Number analyzed (Participants) | 130 | 118
units on a scale | 12.38 (11.23) | 10.96 (11.97)

24. Secondary Outcome: To Compare the Change in SF-12 Physical Health Score From Pre-op to 2 Years Between Sigma RP and Sigma Fixed Treatment Groups in PCL Retaining Arm
Description: as for outcome 23
Time Frame: Change from pre-op to 2 years
Population: Due to consent withdrawals, deaths, lost to follow up, revisions, subjects whose patella were resurfaced, mis-randomized, those who did not wish to continue in the study, and incomplete or unavailable assessments, 139 subjects in the PFC Sigma Fixed Bearing and 130 subjects in the PFC Sigma RP Treatment Groups were available for this outcome.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | PFC Sigma Fixed Bearing PCL Retained | PFC Sigma RP PCL Retained
Number analyzed (Participants) | 139 | 130
units on a scale | 10.47 (10.76) | 9.68 (11.38)

25. Secondary Outcome: To Compare the Change in SF-12 Physical Health Score From Pre-op to 5 Years Between Sigma RP and Sigma Fixed Treatment Groups in PCL Sacrificing Arm
Description: as for outcome 23
Time Frame: Change from pre-op to 5 years
Population: Due to consent withdrawals, deaths, lost to follow up, revisions, subjects whose patella were resurfaced, mis-randomized, those who did not wish to continue in the study, and incomplete or unavailable assessments, 107 subjects in the PFC Sigma Fixed Bearing and 109 subjects in the PFC Sigma RP Treatment Groups were available for this outcome.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | PFC Fixed Bearing PCL Sacrificed | PFC Sigma RP PCL Sacrificed
Number analyzed (Participants) | 107 | 109
units on a scale | 10.90 (11.84) | 8.75 (12.47)

26. Secondary Outcome: To Compare the Change in SF-12 Mental Health Score From Pre-op to 2 Years Between Sigma RP and Sigma Fixed Treatment Groups in PCL Sacrificing Arm
Description: as for outcome 23
Time Frame: Change from pre-op to 2 years
Population: as for outcome 23
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | PFC Fixed Bearing PCL Sacrificed | PFC Sigma RP PCL Sacrificed
Number analyzed (Participants) | 130 | 118
units on a scale | 0.67 (10.71) | 1.91 (10.27)

27. Secondary Outcome: To Compare the Change in SF-12 Mental Health Score From Pre-op to 2 Years Between Sigma RP and Sigma Fixed Treatment Groups in PCL Retaining Arm
Description: as for outcome 23
Time Frame: Change from pre-op to 2 years
Population: as for outcome 24
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | PFC Sigma Fixed Bearing PCL Retained | PFC Sigma RP PCL Retained
Number analyzed (Participants) | 139 | 130
units on a scale | 1.86 (12.69) | 0.26 (11.86)

28. Secondary Outcome: To Compare the Change in SF-12 Mental Health Score From Pre-op to 5 Years Between Sigma RP and Sigma Fixed Treatment Groups in PCL Sacrificing Arm
Description: as for outcome 23
Time Frame: Change from pre-op to 5 years
Population: as for outcome 25
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | PFC Fixed Bearing PCL Sacrificed | PFC Sigma RP PCL Sacrificed
Number analyzed (Participants) | 107 | 109
units on a scale | 1.51 (12.74) | 1.98 (10.64)

29. Secondary Outcome: To Compare the Change in Patella Score From Pre-op to 2 Years Between Sigma RP and Sigma Fixed Treatment Groups in PCL Sacrificing Arm
Description: The Patella Score is completed by the clinicians and assesses the anterior knee pain, quadriceps strength, ability to rise from a chair and stair climbing. The Patella Score ranges from 3 to 30 points with higher scores indicating better functionality and lower scores indicating poorer functionality.
Time Frame: Change from pre-op to 2 years
Population: Due to consent withdrawals, deaths, lost to follow up, revisions, subjects whose patella were resurfaced, mis-randomized, those who did not wish to continue in the study, and incomplete or unavailable assessments, 152 subjects in the PFC Sigma Fixed Bearing and 141 subjects in the PFC Sigma RP Treatment Groups were available for this outcome.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | PFC Fixed Bearing PCL Sacrificed | PFC Sigma RP PCL Sacrificed
Number analyzed (Participants) | 152 | 141
units on a scale | 9.6 (6.89) | 8.4 (7.40)

30. Secondary Outcome: To Compare the Change in Patella Score From Pre-op to 2 Years Between Sigma RP and Sigma Fixed Treatment Groups in PCL Retaining Arm
Description: as for outcome 29
Time Frame: Change from pre-op to 2 years
Population: Due to consent withdrawals, deaths, lost to follow up, revisions, subjects whose patella were resurfaced, mis-randomized, those who did not wish to continue in the study, and incomplete or unavailable assessments, 153 subjects in the PFC Sigma Fixed Bearing and 144 subjects in the PFC Sigma RP Treatment Groups were available for this outcome.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | PFC Sigma Fixed Bearing PCL Retained | PFC Sigma RP PCL Retained
Number analyzed (Participants) | 153 | 144
units on a scale | 10.6 (7.14) | 9.7 (7.35)

31. Secondary Outcome: To Compare the Change in Patella Score From Pre-op to 5 Years Between Sigma RP and Sigma Fixed Treatment Groups in PCL Sacrificing Arm
Description: as for outcome 29
Time Frame: Change from pre-op to 5 years
Population: Due to consent withdrawals, deaths, lost to follow up, revisions, subjects whose patella were resurfaced, mis-randomized, those who did not wish to continue in the study, and incomplete or unavailable assessments, 122 subjects in the PFC Sigma Fixed Bearing and 122 subjects in the PFC Sigma RP Treatment Groups were available for this outcome.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | PFC Fixed Bearing PCL Sacrificed | PFC Sigma RP PCL Sacrificed
Number analyzed (Participants) | 122 | 122
units on a scale | 10.0 (7.04) | 8.6 (8.07)

32. Secondary Outcome: To Compare the Percentage of Subjects With at Least 1 Tibial Radiolucency Between Sigma RP and Sigma Fixed Treatment Groups in PCL Sacrificing Arm
Description: Tibial Radiolucency observes a radiolucent line (of 0.5mm or wider) on the radiograph around the tibial component.
Time Frame: 2 years
Population: as for outcome 17
Measure: Number; unit: percentage of participants
Arm/Group | PFC Fixed Bearing PCL Sacrificed | PFC Sigma RP PCL Sacrificed
Number analyzed (Participants) | 176 | 176
percentage of participants | 9 | 14

33. Secondary Outcome: To Compare the Percentage of Subjects With at Least 1 Tibial Radiolucency Between Sigma RP and Sigma Fixed Treatment Groups in PCL Retaining Arm
Description: Tibial Radiolucency observes a radiolucent line (of 0.5mm or wider) on the radiograph around the tibial component.
Time Frame: 2 years
Population: as for outcome 6
Measure: Number; unit: percentage of participants
Arm/Group | PFC Sigma Fixed Bearing PCL Retained | PFC Sigma RP PCL Retained
Number analyzed (Participants) | 170 | 161
percentage of participants | 9 | 20

34. Secondary Outcome: To Compare the Percentage of Subjects With at Least 1 Tibial Radiolucency Between Sigma RP and Sigma Fixed Treatment Groups in PCL Sacrificing Arm
Description: Tibial Radiolucency observes a radiolucent line (of 0.5mm or wider) on the radiograph around the tibial component.
Time Frame: 5 Years
Population: as for outcome 17
Measure: Number; unit: percentage of participants
Arm/Group | PFC Fixed Bearing PCL Sacrificed | PFC Sigma RP PCL Sacrificed
Number analyzed (Participants) | 176 | 176
percentage of participants | 8 | 6

35. Secondary Outcome: To Compare the Percentage of Subjects With Lateral Release Between Sigma RP and Sigma Fixed Treatment Groups in PCL Sacrificing Arm
Description: Lateral release is a surgical procedure to release tight capsular structures (lateral retinaculum) on the outside of the kneecap (patella). It is performed during knee surgery and allows the kneecap to move smoothly in the center of the knee. Rate information was collected at time of study surgery.
Time Frame: Operative
Population: as for outcome 17
Measure: Number; unit: percentage of participants
Arm/Group | PFC Fixed Bearing PCL Sacrificed | PFC Sigma RP PCL Sacrificed
Number analyzed (Participants) | 176 | 176
percentage of participants | 10 | 10

36. Secondary Outcome: To Compare the Percentage of Subjects With Lateral Release Between Sigma RP and Sigma Fixed Treatment Groups in PCL Retaining Arm
Description: as for outcome 35
Time Frame: Operative
Population: as for outcome 6
Measure: Number; unit: percentage of participants
Arm/Group | PFC Sigma Fixed Bearing PCL Retained | PFC Sigma RP PCL Retained
Number analyzed (Participants) | 170 | 161
percentage of participants | 7 | 7

37. Secondary Outcome: To Compare the Survivorship Analysis Results Between Sigma RP and Sigma Fixed Treatment Groups in PCL Sacrificing Arm
Description: Kaplan Meier survivorship analysis estimates the proportion of a population that will survive past a certain time avoiding a certain event. In this study, the event is removal of any component for any reason, also known as revision for any reason. Survival estimates are provided when 40 devices are left still being followed.
Time Frame: 2 Years
Population: as for outcome 17
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | PFC Fixed Bearing PCL Sacrificed | PFC Sigma RP PCL Sacrificed
Number analyzed (Participants) | 176 | 176
percentage of participants | 98.9 [95.5 to 99.7] | 98.3 [94.7 to 99.4]

38. Secondary Outcome: To Compare the Survivorship Analysis Results Between Sigma RP and Sigma Fixed Treatment Groups in PCL Retaining Arm
Description: as for outcome 37
Time Frame: 2 Years
Population: as for outcome 6
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | PFC Sigma Fixed Bearing PCL Retained | PFC Sigma RP PCL Retained
Number analyzed (Participants) | 170 | 161
percentage of participants | 99.4 [95.9 to 99.9] | 98.1 [94.3 to 99.4]

39. Secondary Outcome: To Compare the Survivorship Analysis Results Between Sigma RP and Sigma Fixed Treatment Groups in PCL Sacrificing Arm
Description: as for outcome 37
Time Frame: 5 Years
Population: as for outcome 17
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | PFC Fixed Bearing PCL Sacrificed | PFC Sigma RP PCL Sacrificed
Number analyzed (Participants) | 176 | 176
percentage of participants | 96.3 [92.0 to 98.3] | 97.6 [93.7 to 99.1]

40. Secondary Outcome: To Compare the Percentage of Subjects With No Anterior Knee Pain Between Sigma RP and Sigma Fixed Bearing Treatment Groups With Patella Resurfacing in the PCL Sacrificing Arm
Description: as for outcome 17
Time Frame: 2 Years
Population: Due to consent withdrawals, deaths, lost to follow up, revisions, subjects whose patella were resurfaced, mis-randomized, those who did not wish to continue in the study, and incomplete or unavailable assessments, 88 subjects in the PFC Sigma Fixed Bearing and 89 subjects in the PFC Sigma RP Treatment Groups were available for this outcome.
Measure: Number; unit: percentage of participants
Arm/Group | PFC Fixed Bearing PCL Sacrificed | PFC Sigma RP PCL Sacrificed
Number analyzed (Participants) | 88 | 89
percentage of participants | 75 | 69

41. Secondary Outcome: To Compare the Percentage of Subjects With No Anterior Knee Pain Between Sigma RP and Sigma Fixed Bearing Treatment Groups Without Patella Resurfacing in the PCL Sacrificing Arm
Description: as for outcome 17
Time Frame: 2 Years
Population: Due to consent withdrawals, deaths, lost to follow up, revisions, subjects whose patella were resurfaced, mis-randomized, those who did not wish to continue in the study, and incomplete or unavailable assessments, 88 subjects in the PFC Sigma Fixed Bearing and 87 subjects in the PFC Sigma RP Treatment Groups were available for this outcome.
Measure: Number; unit: percentage of participants
Arm/Group | PFC Fixed Bearing PCL Sacrificed | PFC Sigma RP PCL Sacrificed
Number analyzed (Participants) | 88 | 87
percentage of participants | 72 | 66

42. Secondary Outcome: To Compare the Percentage of Subjects With No Anterior Knee Pain Between Sigma RP and Sigma Fixed Bearing Treatment Groups With Patella Resurfacing in the PCL Sacrificing Arm
Description: as for outcome 17
Time Frame: 5 Years
Population: as for outcome 40
Measure: Number; unit: percentage of participants
Arm/Group | PFC Fixed Bearing PCL Sacrificed | PFC Sigma RP PCL Sacrificed
Number analyzed (Participants) | 88 | 89
percentage of participants | 65 | 54

43. Secondary Outcome: To Compare the Percentage of Subjects With No Anterior Knee Pain Between Sigma RP and Sigma Fixed Bearing Treatment Groups Without Patella Resurfacing in the PCL Sacrificing Arm
Description: as for outcome 17
Time Frame: 5 Years
Population: as for outcome 41
Measure: Number; unit: percentage of participants
Arm/Group | PFC Fixed Bearing PCL Sacrificed | PFC Sigma RP PCL Sacrificed
Number analyzed (Participants) | 88 | 87
percentage of participants | 57 | 53

44. Secondary Outcome: To Compare the Percentage of Subjects With Good Quadriceps Strength Between Sigma RP and Sigma Fixed Bearing Treatment Groups With Patella Resurfacing in the PCL Sacrificing Arm
Description: as for outcome 20
Time Frame: 2 Years
Population: as for outcome 40
Measure: Number; unit: percentage of participants
Arm/Group | PFC Fixed Bearing PCL Sacrificed | PFC Sigma RP PCL Sacrificed
Number analyzed (Participants) | 88 | 89
percentage of participants | 88 | 83

45. Secondary Outcome: To Compare the Percentage of Subjects With Good Quadriceps Strength Between Sigma RP and Sigma Fixed Bearing Treatment Groups Without Patella Resurfacing in the PCL Sacrificing Arm
Description: as for outcome 20
Time Frame: 2 Years
Population: as for outcome 41
Measure: Number; unit: percentage of participants
Arm/Group | PFC Fixed Bearing PCL Sacrificed | PFC Sigma RP PCL Sacrificed
Number analyzed (Participants) | 88 | 87
percentage of participants | 88 | 86

46. Secondary Outcome: To Compare the Percentage of Subjects With Good Quadriceps Strength Between Sigma RP and Sigma Fixed Bearing Treatment Groups With Patella Resurfacing in the PCL Sacrificing Arm
Description: as for outcome 20
Time Frame: 5 Years
Population: as for outcome 40
Measure: Number; unit: percentage of participants
Arm/Group | PFC Fixed Bearing PCL Sacrificed | PFC Sigma RP PCL Sacrificed
Number analyzed (Participants) | 88 | 89
percentage of participants | 65 | 71

47. Secondary Outcome: To Compare the Percentage of Subjects With Good Quadriceps Strength Between Sigma RP and Sigma Fixed Bearing Treatment Groups Without Patella Resurfacing in the PCL Sacrificing Arm
Description: as for outcome 20
Time Frame: 5 Years
Population: as for outcome 41
Measure: Number; unit: percentage of participants
Arm/Group | PFC Fixed Bearing PCL Sacrificed | PFC Sigma RP PCL Sacrificed
Number analyzed (Participants) | 88 | 87
percentage of participants | 66 | 64

48. Secondary Outcome: To Compare the Change in Patella Score From Pre-op to 2 Years Between Sigma RP and Sigma Fixed Bearing Treatment Groups With Patella Resurfacing in the PCL Sacrificing Arm
Description: as for outcome 29
Time Frame: Change from pre-op to 2 years
Population: Due to consent withdrawals, deaths, lost to follow up, revisions, subjects whose patella were resurfaced, mis-randomized, those who did not wish to continue in the study, and incomplete or unavailable assessments, 75 subjects in the PFC Sigma Fixed Bearing and 71 subjects in the PFC Sigma RP Treatment Groups were available for this outcome.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | PFC Fixed Bearing PCL Sacrificed | PFC Sigma RP PCL Sacrificed
Number analyzed (Participants) | 75 | 71
units on a scale | 8.8 (7.03) | 9.4 (6.37)

49. Secondary Outcome: To Compare the Change in Patella Score From Pre-op to 2 Years Between Sigma RP and Sigma Fixed Bearing Treatment Groups Without Patella Resurfacing in the PCL Sacrificing Arm
Description: as for outcome 29
Time Frame: Change from pre-op to 2 years
Population: Due to consent withdrawals, deaths, lost to follow up, revisions, subjects whose patella were resurfaced, mis-randomized, those who did not wish to continue in the study, and incomplete or unavailable assessments, 77 subjects in the PFC Sigma Fixed Bearing and 70 subjects in the PFC Sigma RP Treatment Groups were available for this outcome.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | PFC Fixed Bearing PCL Sacrificed | PFC Sigma RP PCL Sacrificed
Number analyzed (Participants) | 77 | 70
units on a scale | 10.3 (6.72) | 7.5 (8.25)

50. Secondary Outcome: To Compare the Change in Patella Score From Pre-op to 5 Years Between Sigma RP and Sigma Fixed Bearing Treatment Groups With Patella Resurfacing in the PCL Sacrificing Arm
Description: as for outcome 29
Time Frame: Change from pre-op to 5 years
Population: Due to consent withdrawals, deaths, lost to follow up, revisions, subjects whose patella were resurfaced, mis-randomized, those who did not wish to continue in the study, and incomplete or unavailable assessments, 60 subjects in the PFC Sigma Fixed Bearing and 62 subjects in the PFC Sigma RP Treatment Groups were available for this outcome.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | PFC Fixed Bearing PCL Sacrificed | PFC Sigma RP PCL Sacrificed
Number analyzed (Participants) | 60 | 62
units on a scale | 8.9 (7.35) | 9.1 (7.16)

51. Secondary Outcome: To Compare the Change in Patella Score From Pre-op to 5 Years Between Sigma RP and Sigma Fixed Bearing Treatment Groups Without Patella Resurfacing in the PCL Sacrificing Arm
Description: as for outcome 29
Time Frame: Change from pre-op to 5 years
Population: Due to consent withdrawals, deaths, lost to follow up, revisions, subjects whose patella were resurfaced, mis-randomized, those who did not wish to continue in the study, and incomplete or unavailable assessments, 62 subjects in the PFC Sigma Fixed Bearing and 60 subjects in the PFC Sigma RP Treatment Groups were available for this outcome.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | PFC Fixed Bearing PCL Sacrificed | PFC Sigma RP PCL Sacrificed
Number analyzed (Participants) | 62 | 60
units on a scale | 11.2 (6.57) | 8.1 (8.94)

ADVERSE EVENTS:
Arm/Group | PFC Fixed Bearing PCL Sacrificed | PFC Sigma RP PCL Sacrificed | PFC Sigma Fixed Bearing PCL Retained | PFC Sigma RP PCL Retained
Serious Adverse Events (participants affected / at risk) | 111/193 | 107/196 | 110/170 | 96/161
Other Adverse Events (participants affected / at risk) | 0/193 | 0/196 | 0/170 | 0/161
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | PFC Fixed Bearing PCL Sacrificed (N=193) | PFC Sigma RP PCL Sacrificed (N=196) | PFC Sigma Fixed Bearing PCL Retained (N=170) | PFC Sigma RP PCL Retained (N=161)
Anaemia (Blood and lymphatic system disorders) | 1 | 2 | 0 | 0
Iron deficiency anaemia (Blood and lymphatic system disorders) | 0 | 0 | 1 | 0
Lymphocytosis (Blood and lymphatic system disorders) | 1 | 0 | 0 | 0
Angina pectoris (Cardiac disorders) | 2 | 4 | 2 | 1
Arrhythmia (Cardiac disorders) | 1 | 0 | 0 | 0
Atrial fibrillation (Cardiac disorders) | 3 | 2 | 2 | 4
Atrial flutter (Cardiac disorders) | 0 | 1 | 1 | 0
Atrioventricular block (Cardiac disorders) | 0 | 0 | 2 | 0
Atrioventricular block complete (Cardiac disorders) | 1 | 0 | 0 | 0
Cardiac arrest (Cardiac disorders) | 0 | 2 | 1 | 0
Cardiac failure (Cardiac disorders) | 1 | 3 | 0 | 1
Cardiac disorders NEC (Cardiac disorders) | 0 | 0 | 1 | 0
Cardiovascular disorder (Cardiac disorders) | 1 | 2 | 1 | 1
Coronary artery disease (Cardiac disorders) | 0 | 2 | 1 | 4
Heart enlarged (Cardiac disorders) | 0 | 1 | 0 | 0
Mitral valve incompetence (Cardiac disorders) | 0 | 1 | 1 | 0
Myocardial infarction (Cardiac disorders) | 2 | 4 | 2 | 0
Tinnitus (Ear and labyrinth disorders) | 0 | 0 | 0 | 1
Blindness (Eye disorders) | 1 | 1 | 0 | 1
Cataract (Eye disorders) | 2 | 0 | 10 | 4
Eye haemorrhage (Eye disorders) | 0 | 1 | 0 | 0
Diplopia (Eye disorders) | 0 | 0 | 1 | 0
Glaucoma (Eye disorders) | 0 | 0 | 2 | 0
Macular degeneration (Eye disorders) | 0 | 0 | 1 | 0
Macular hole (Eye disorders) | 0 | 0 | 0 | 1
Uveitis (Eye disorders) | 0 | 0 | 0 | 1
Visual acuity reduced (Eye disorders) | 0 | 0 | 1 | 0
Abdominal discomfort (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Abdominal mass (Gastrointestinal disorders) | 1 | 1 | 0 | 0
Abdominal pain (Gastrointestinal disorders) | 2 | 2 | 2 | 2
Abdominal pain upper (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Anal haemorrhage (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Diarrhoea (Gastrointestinal disorders) | 2 | 0 | 0 | 1
Ascites (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Dyspepsia (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Constipation (Gastrointestinal disorders) | 0 | 0 | 1 | 2
Faeces discoloured (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Faecal incontinence (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Faeces pale (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Haemorrhoidal haemorrhage (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Frequent bowel movements (Gastrointestinal disorders) | 2 | 0 | 0 | 0
Hiatal hernia (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Gastric ulcer (Gastrointestinal disorders) | 1 | 1 | 0 | 0
Hiatus hernia (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Haematemesis (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Inguinal hernia (Gastrointestinal disorders) | 1 | 1 | 0 | 0
Intestinal perforation (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Obstruction gastric (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Oral pain (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Pancreatitis acute (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Rectal haemorrhage (Gastrointestinal disorders) | 2 | 0 | 0 | 1
Umbilical hernia (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Chest pain (General disorders) | 3 | 3 | 0 | 0
Death- Unknown (General disorders) | 16 | 11 | 3 | 3
Device connection issue (General disorders) | 0 | 1 | 0 | 0
Device dislocation (General disorders) | 0 | 2 | 1 | 0
Device extrusion (General disorders) | 0 | 1 | 0 | 0
Gait disturbance (General disorders) | 1 | 0 | 0 | 0
Malaise (General disorders) | 0 | 1 | 0 | 0
Medical device complication (General disorders) | 1 | 0 | 0 | 0
Pain (General disorders) | 4 | 1 | 1 | 2
Spinal pain (General disorders) | 1 | 0 | 0 | 0
Weight bearing difficulty (General disorders) | 0 | 1 | 0 | 0
Chest discomfort (General disorders) | 0 | 0 | 1 | 0
Device component issue (General disorders) | 0 | 0 | 0 | 1
Device failure (General disorders) | 0 | 0 | 0 | 1
Hernia (General disorders) | 0 | 0 | 1 | 1
Oedema peripheral (General disorders) | 0 | 0 | 1 | 1
Pain and discomfort NEC (General disorders) | 0 | 0 | 3 | 0
Pyrexia (General disorders) | 0 | 0 | 0 | 1
Surgical failure (General disorders) | 0 | 0 | 1 | 0
Swelling (General disorders) | 0 | 0 | 3 | 1
Cholelithiasis (Hepatobiliary disorders) | 3 | 0 | 0 | 1
Biliary colic (Hepatobiliary disorders) | 1 | 0 | 0 | 0
Cholecystitis (Hepatobiliary disorders) | 0 | 1 | 0 | 0
Cholecystitis chronic (Hepatobiliary disorders) | 1 | 0 | 0 | 0
Gallbladder perforation (Hepatobiliary disorders) | 1 | 1 | 0 | 0
Jaundice (Hepatobiliary disorders) | 0 | 2 | 0 | 0
Cellulitis (Infections and infestations) | 1 | 0 | 0 | 0
Diverticulitis (Infections and infestations) | 2 | 0 | 1 | 1
Helicobacter gastritis (Infections and infestations) | 0 | 1 | 0 | 0
Implant site infection (Infections and infestations) | 1 | 0 | 0 | 0
Infection (Infections and infestations) | 1 | 2 | 2 | 1
Lower respiratory tract infection (Infections and infestations) | 1 | 1 | 1 | 2
Peritonitis (Infections and infestations) | 1 | 0 | 0 | 0
Pneumonia (Infections and infestations) | 0 | 3 | 1 | 2
Post procedural infection (Infections and infestations) | 1 | 0 | 2 | 0
Postoperative wound infection (Infections and infestations) | 0 | 1 | 0 | 0
Sepsis (Infections and infestations) | 0 | 1 | 1 | 0
Staphylococcal infection (Infections and infestations) | 3 | 2 | 0 | 3
Stitch abscess (Infections and infestations) | 1 | 0 | 0 | 0
Streptococcal infection (Infections and infestations) | 1 | 0 | 1 | 0
Tuberculosis (Infections and infestations) | 1 | 0 | 0 | 0
Urinary tract infection (Infections and infestations) | 1 | 0 | 1 | 2
Wound infection (Infections and infestations) | 2 | 2 | 1 | 2
Wound infection staphylococcal (Infections and infestations) | 0 | 1 | 0 | 0
Clostridium difficile colitis (Infections and infestations) | 0 | 0 | 1 | 0
Clostridium difficile infection (Infections and infestations) | 0 | 0 | 0 | 1
Ear infection staphylococcal (Infections and infestations) | 0 | 0 | 1 | 0
Gastroenteritis (Infections and infestations) | 0 | 0 | 1 | 0
Helicobacter infection (Infections and infestations) | 0 | 0 | 0 | 1
Infected dermal cyst (Infections and infestations) | 0 | 0 | 0 | 1
Lobar pneumonia (Infections and infestations) | 0 | 0 | 0 | 1
Lower respiratory tract infections NEC (Infections and infestations) | 0 | 0 | 1 | 0
Osteomyelitis (Infections and infestations) | 0 | 0 | 2 | 0
Pneumonia legionella (Infections and infestations) | 0 | 0 | 1 | 0
Ankle fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0
Cervical vertebral fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1
Concussion (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0
Ear injury (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1
Facial bones fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0
Fall (Injury, poisoning and procedural complications) | 5 | 8 | 4 | 7
Femoral neck fracture (Injury, poisoning and procedural complications) | 3 | 0 | 4 | 1
Femur fracture (Injury, poisoning and procedural complications) | 0 | 1 | 1 | 1
Glaucoma traumatic (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1
Head injury (Injury, poisoning and procedural complications) | 2 | 0 | 1 | 0
Hip fracture (Injury, poisoning and procedural complications) | 0 | 1 | 1 | 0
Humerus fracture (Injury, poisoning and procedural complications) | 1 | 0 | 1 | 0
Joint dislocation (Injury, poisoning and procedural complications) | 2 | 3 | 3 | 1
Joint dislocation postoperative (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1
Joint injury (Injury, poisoning and procedural complications) | 0 | 1 | 1 | 1
Laceration (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1
Ligament rupture (Injury, poisoning and procedural complications) | 0 | 0 | 2 | 1
Limb injury (Injury, poisoning and procedural complications) | 1 | 0 | 1 | 0
Lower limb fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0
Overdose (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1
Pelvic fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0
Radius fracture (Injury, poisoning and procedural complications) | 1 | 0 | 3 | 1
Subdural haemorrhage (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0
Tibia fracture (Injury, poisoning and procedural complications) | 2 | 0 | 0 | 1
Wound complication (Injury, poisoning and procedural complications) | 2 | 2 | 0 | 2
Wound dehiscence (Injury, poisoning and procedural complications) | 0 | 0 | 2 | 0
Wound secretion (Injury, poisoning and procedural complications) | 0 | 1 | 1 | 0
Wrist fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1
Back injury (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Fractured olecranon (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Hand fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0
Post procedural complication (Injury, poisoning and procedural complications) | 1 | 1 | 0 | 0
Post procedural myocardial infarction (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0
Post-traumatic neck syndrome (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Road traffic accident (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Skin wound (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Upper limb fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Bone scan (Investigations) | 1 | 0 | 0 | 0
Endoscopy (Investigations) | 1 | 0 | 0 | 0
Gastrointestinal examination (Investigations) | 0 | 1 | 0 | 0
Haemoglobin decreased (Investigations) | 0 | 1 | 0 | 0
Prostatic specific antigen increased (Investigations) | 0 | 1 | 0 | 0
Staphylococcus test positive (Investigations) | 1 | 1 | 0 | 0
Weight decreased (Investigations) | 0 | 1 | 0 | 0
Chest X-ray abnormal (Investigations) | 0 | 0 | 0 | 2
Computerised tomogram abnormal (Investigations) | 0 | 0 | 0 | 1
Investigation (Investigations) | 0 | 0 | 0 | 1
Liver function test abnormal (Investigations) | 0 | 0 | 0 | 1
Macular reflex abnormal (Investigations) | 0 | 0 | 0 | 1
Weight loss (Investigations) | 0 | 0 | 1 | 1
Decreased appetite (Metabolism and nutrition disorders) | 0 | 1 | 0 | 1
Dehydration (Metabolism and nutrition disorders) | 0 | 0 | 1 | 1
Diabetes mellitus (Metabolism and nutrition disorders) | 2 | 0 | 1 | 2
Type 2 diabetes mellitus (Metabolism and nutrition disorders) | 1 | 2 | 0 | 2
Haemochromatosis (Metabolism and nutrition disorders) | 0 | 2 | 0 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 6 | 7 | 8 | 10
Arthropathy (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 3 | 1 | 1 | 3
Foot deformity (Musculoskeletal and connective tissue disorders) | 1 | 1 | 0 | 1
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1
Joint crepitation (Musculoskeletal and connective tissue disorders) | 0 | 1 | 1 | 0
Joint range of motion decreased (Musculoskeletal and connective tissue disorders) | 1 | 0 | 4 | 2
Joint swelling (Musculoskeletal and connective tissue disorders) | 2 | 4 | 1 | 0
Limb discomfort (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1
Lumbar spinal stenosis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0
Mobility decreased (Musculoskeletal and connective tissue disorders) | 1 | 2 | 0 | 1
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 2 | 0
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 27 | 28 | 36 | 23
Osteonecrosis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1
Pain groin (Musculoskeletal and connective tissue disorders) | 1 | 2 | 0 | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 2 | 1 | 0 | 1
Patellofemoral pain syndrome (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1
Periarthritis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0
Rheumatoid arthritis (Musculoskeletal and connective tissue disorders) | 1 | 1 | 0 | 1
Rotator cuff syndrome (Musculoskeletal and connective tissue disorders) | 0 | 2 | 1 | 0
Spinal column stenosis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1
Stiff knees (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1
Arthritis (Musculoskeletal and connective tissue disorders) | 1 | 1 | 0 | 0
Back disorder (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0
Dupuytren's contracture (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0
Haemarthrosis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0
Joint contracture (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0
Joint instability (Musculoskeletal and connective tissue disorders) | 1 | 2 | 0 | 0
Joint lock (Musculoskeletal and connective tissue disorders) | 1 | 1 | 0 | 0
Joint stiffness (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0
Low back pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0
Muscular weakness (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0
Musculoskeletal deformity (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0
Musculoskeletal stiffness (Musculoskeletal and connective tissue disorders) | 3 | 0 | 0 | 0
Osteosclerosis (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0
Pain in elbow (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0
Pain in hand (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0
Scoliosis (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0
Synovitis (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0
Toe osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0
Ataxia (Nervous system disorders) | 0 | 0 | 0 | 1
Carpal tunnel syndrome (Nervous system disorders) | 2 | 0 | 4 | 2
Cerebral haemorrhage (Nervous system disorders) | 0 | 0 | 1 | 0
Cerebral infarction (Nervous system disorders) | 0 | 1 | 1 | 0
Cerebrovascular accident (Nervous system disorders) | 5 | 2 | 2 | 4
Convulsion (Nervous system disorders) | 0 | 0 | 0 | 1
Dementia (Nervous system disorders) | 2 | 2 | 1 | 1
Dementia Alzheimer's type (Nervous system disorders) | 1 | 0 | 2 | 0
Headache (Nervous system disorders) | 0 | 0 | 0 | 1
Hemiparesis (Nervous system disorders) | 1 | 1 | 1 | 1
Radial nerve palsy (Nervous system disorders) | 0 | 0 | 1 | 0
Sciatica (Nervous system disorders) | 0 | 0 | 1 | 0
Sensory loss (Nervous system disorders) | 0 | 0 | 1 | 0
Syncope (Nervous system disorders) | 0 | 0 | 1 | 1
Tethered cord syndrome (Nervous system disorders) | 0 | 0 | 0 | 1
Transient ischaemic attack (Nervous system disorders) | 0 | 0 | 2 | 1
Brain hypoxia (Nervous system disorders) | 0 | 1 | 0 | 0
Burning sensation (Nervous system disorders) | 0 | 1 | 0 | 0
Carotid artery stenosis (Nervous system disorders) | 0 | 1 | 0 | 0
Dizziness (Nervous system disorders) | 2 | 1 | 0 | 0
Dysgraphia (Nervous system disorders) | 1 | 0 | 0 | 0
Hydrocephalus (Nervous system disorders) | 1 | 0 | 0 | 0
Loss of consciousness (Nervous system disorders) | 0 | 1 | 0 | 0
Paraesthesia (Nervous system disorders) | 0 | 1 | 0 | 0
Parkinson's disease (Nervous system disorders) | 0 | 1 | 0 | 0
Sensory disturbance (Nervous system disorders) | 1 | 2 | 0 | 0
Anxiety (Psychiatric disorders) | 0 | 0 | 1 | 0
Confusional state (Psychiatric disorders) | 1 | 0 | 0 | 1
Depression (Psychiatric disorders) | 0 | 0 | 1 | 1
Hallucination, auditory (Psychiatric disorders) | 0 | 0 | 0 | 1
Agitation (Psychiatric disorders) | 1 | 0 | 0 | 0
Completed suicide (Psychiatric disorders) | 1 | 0 | 0 | 0
Haematuria (Renal and urinary disorders) | 1 | 2 | 0 | 1
Renal failure (Renal and urinary disorders) | 0 | 0 | 2 | 1
Renal failure acute (Renal and urinary disorders) | 0 | 0 | 0 | 1
Renal failure chronic (Renal and urinary disorders) | 0 | 2 | 1 | 0
Renal mass (Renal and urinary disorders) | 0 | 0 | 0 | 1
Chromaturia (Renal and urinary disorders) | 0 | 1 | 0 | 0
Incontinence (Renal and urinary disorders) | 2 | 0 | 0 | 0
Micturition urgency (Renal and urinary disorders) | 1 | 0 | 0 | 0
Nephrolithiasis (Renal and urinary disorders) | 0 | 3 | 0 | 0
Urinary retention (Renal and urinary disorders) | 2 | 0 | 0 | 0
Urine flow decreased (Renal and urinary disorders) | 0 | 1 | 0 | 0
Breast mass (Reproductive system and breast disorders) | 0 | 1 | 0 | 1
Testicular swelling (Reproductive system and breast disorders) | 1 | 0 | 0 | 0
Cystocele (Reproductive system and breast disorders) | 0 | 0 | 0 | 1
Postmenopausal haemorrhage (Reproductive system and breast disorders) | 0 | 0 | 2 | 0
Vaginal prolapse (Reproductive system and breast disorders) | 0 | 0 | 1 | 2
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 4 | 4 | 0 | 3
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 3 | 3 | 1 | 2
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1
Sleep apnoea syndrome (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1
Throat pain (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0
Tonsillar disorder (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0
Emphysema (Respiratory, thoracic and mediastinal disorders) | 0 | 2 | 0 | 0
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0
Interstitial lung disease (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 0 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0
Respiratory disorder (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0
Hyperkeratosis (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0
Angioplasty (Surgical and medical procedures) | 0 | 1 | 0 | 0
Ankle arthroplasty (Surgical and medical procedures) | 0 | 1 | 0 | 0
Cholecystectomy (Surgical and medical procedures) | 0 | 1 | 1 | 0
Hip arthroplasty (Surgical and medical procedures) | 1 | 1 | 0 | 1
Hospitalisation (Surgical and medical procedures) | 3 | 5 | 3 | 5
Joint arthroplasty (Surgical and medical procedures) | 1 | 2 | 0 | 0
Knee arthroplasty (Surgical and medical procedures) | 12 | 11 | 4 | 1
Rotator cuff repair (Surgical and medical procedures) | 0 | 1 | 0 | 0
Shoulder operation (Surgical and medical procedures) | 1 | 0 | 0 | 0
Wound drainage (Surgical and medical procedures) | 1 | 0 | 0 | 0
Cellulitis (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1
Skin lesion (Skin and subcutaneous tissue disorders) | 0 | 0 | 2 | 0
Skin ulcer (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 1
Breast lump removal (Surgical and medical procedures) | 0 | 0 | 0 | 1
Hysterectomy (Surgical and medical procedures) | 0 | 0 | 1 | 0
Leg amputation (Surgical and medical procedures) | 0 | 0 | 1 | 0
Surgery (Surgical and medical procedures) | 0 | 0 | 1 | 0
Aortic aneurysm (Vascular disorders) | 0 | 0 | 1 | 1
Aortic aneurysm rupture (Vascular disorders) | 0 | 0 | 1 | 0
Deep vein thrombosis (Vascular disorders) | 4 | 7 | 2 | 3
Haemorrhage (Vascular disorders) | 0 | 0 | 1 | 1
Orthostatic hypotension (Vascular disorders) | 0 | 0 | 0 | 2
Peripheral artery aneurysm (Vascular disorders) | 0 | 0 | 0 | 1
Varicose vein (Vascular disorders) | 0 | 0 | 2 | 0
Embolism (Vascular disorders) | 1 | 0 | 0 | 0
Haematoma (Vascular disorders) | 2 | 0 | 0 | 0
Peripheral vascular disorder (Vascular disorders) | 1 | 0 | 0 | 0
Phlebitis (Vascular disorders) | 0 | 1 | 0 | 0
Post thrombotic syndrome (Vascular disorders) | 0 | 1 | 0 | 0
Adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1 | 4 | 2
Benign neoplasm of bladder (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0
Bladder cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1 | 0 | 0
Bladder neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0
Bladder neoplasms (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1 | 1 | 3
Hepatic cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0
Invasive ductal breast carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0
Lung metastases (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0
Lung neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 2 | 3 | 0
Malignant melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 1 | 0
Metastases to bone (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0
Neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 1 | 0 | 0
Non-Hodgkin's lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 1
Oesophageal adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0
Pelvic neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1 | 1 | 2
Prostate cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 2 | 0 | 0
Prostatic neoplasms malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 2 | 0 | 0
Small intestine adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0
Uterine cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0
Benign renal neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1
Brain secondaries (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0
Gastrointestinal carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 2
Lipoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0
Lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 2 | 0
Meningioma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0
Metastases to central nervous system (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1
Metastasis (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1
Ovarian cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1
Pituitary tumor NOS (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 1
Rectal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0
Skin cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1
Squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1
Ischaemic Heart Disease (Cardiac disorders) | 0 | 1 | 0 | 0
Cyst (General disorders) | 1 | 0 | 0 | 0
Periorbital contusion (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0
Bone Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0
Gastric Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0
Liver Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0
Oesophageal carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0
Nasal Polyps (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0
Cold Sweat (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
DePuy reserves the right to review the contents of publications in advance.The PI may freely disclose the trial results only after DePuy has been given the opportunity of reviewing the proposed results communications at least 30 days prior to the intended release.DePuy will advise the PI of any perceived errors,omissions or corrections but the PI will retain final editorial control.In case of disagreement,DePuy and the PI will make every effort to meet in order to discuss and resolve any issues.